CLINICAL TRIAL: NCT02346305
Title: Multicenter Prospective and Observational Cohort of Respiratory Failure Patients Treated for the First Time With Non-invasive Ventilation (NIV) at Home
Brief Title: Cohort of Respiratory Failure Patients Treated for the First Time With Non-Invasive Ventilation at Home
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2014 - NIV - 14734
Record Dates: First submitted 2015-01-09; First posted 2015-01-27 (Estimated); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years

INTERVENTIONS:
Device: Non-invasive ventilation — Home NIV installation

SUMMARY:
The effectiveness of NIV is clearly demonstrated but no recent studies describe the prescription based on clinical data and the conditions of using NIV at home according the various respiratory diseases.

The investigators' purpose is that a better knowledge of NIV practices could improve both the quality to support patients at home and the efficacy of the treatment.

The main objective of this study is to analyze the clinical data justifying the prescription of NIV advice according respiratory disease. The secondary objectives are to study comorbidities, treatment failures, survival rate during the study period.

ELIGIBILITY:
Inclusion Criteria:

* No previous experience with domiciliary non-invasive ventilation
* Adult patients, ≥ 18 years of age
* Without tracheotomy
* No evolutive cancer
* No significant psychiatric disease
* Possible medical monitoring

Exclusion Criteria:

* Evolutive cancer
* Inability to understand rationale and/or consent form for study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with respiratoy insufficiency
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2015-01; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Clinical data leading to NIV device prescription | Day 1
  Age, blood gases, BMI, etiology, pulmonary function,comorbidities

SECONDARY OUTCOMES:
Change in blood gases | 4 months, 1 year and 2 years after inclusion
Change in the possible comorbidities | 4 months, 1 year and 2 years after inclusion
Treatment compliance | Initiation of treatment to 4 months
Treatment compliance | 4 months to 1 year
Treatment compliance | 1 year to 2 years (end of study)
Hospitalizations | 4 months
  During the study period all hospitalizations will be notify
Hospitalizations | 1 year
  During the study period all hospitalizations will be notify
Hospitalizations | 2 years
  During the study period all hospitalizations will be notify
Survival rate | 4 months
Survival rate | 1 year
Survival rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Claudio RABEC, MD, Principal Investigator — Centre Hospitalier Universitaire Dijon
Locations (16):
- France (16):
  - CHU d'Angers, Angers
  - CHU de Besançon, Besançon
  - CH de Cannes, Cannes
  - CHU de Dijon, Dijon
  - Garches, Garches
  - CHU de Grenoble, Grenoble
  - CHD de la Réunion, La Réunion
  - CHU de Lille, Lille
  - CHU de Limoges, Limoges
  - CHU de Nancy, Nancy
  - AP-HP Pitié-Salpêtrière, Paris
  - Hôpital Edouard Rist, Paris
  - CHU de Rouen, Rouen
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - Hôpital Robert Schuman, Vantoux